CLINICAL TRIAL: NCT04995523
Title: Phase I/II, Open-label, Dose Escalation and Dose Expansion Study to Evaluate Safety, Pharmacokinetics, Pharmacodynamics and Efficacy of AZD2936 Anti-TIGIT/Anti-PD-1 Bispecific Antibody in Participants With Advanced or Metastatic NSCLC
Brief Title: A Study of AZD2936 Anti-TIGIT/Anti-PD-1 Bispecific Antibody in Participants With Advanced or Metastatic NSCLC
Acronym: ARTEMIDE-01
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D7020C00001; 2023-508262-15-00 (Registry Identifier: EU CT Number); 2021-000857-23 (EudraCT Number)
Record Dates: First submitted 2021-07-16; First posted 2021-08-09 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: TIGIT, Anti-TIGIT; PD-1, Anti-PD-1; NSCLC, Non-small Cell Lung Cancer; Advanced, Metastatic, Solid Tumor, Solid Tumour; Stage 3 NSCLC, Stage III NSCLC; Stage 4 NSCLC, Stage IV NSCLC; PD L1+ tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: The study includes 5 parts: Part A: Dose escalation; B & C & E: Dose expansion non-randomized; D: Randomized RP2D & alternative dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Escalation Part A: Checkpoint inhibitor (CPI) experienced Non-small Cell Lung Cancer (NSCLC) (Experimental): Rilvegostomig Intravenous (IV) monotherapy
  Interventions: Drug: AZD2936
- Dose Expansion Part B: CPI experienced NSCLC (Experimental): Rilvegostomig IV monotherapy
  Interventions: Drug: AZD2936
- Dose Expansion Part C: CPI Naive NSCLC (Experimental): Rilvegostomig IV monotherapy
  Interventions: Drug: AZD2936
- Dose Expansion Part D: CPI Naive NSCLC (Experimental): Rilvegostomig IV monotherapy
  Interventions: Drug: AZD2936
- Dose Expansion Part E: treatment Naive Squamous NSCLC (Experimental): Rilvegostomig IV monotherapy
  Interventions: Drug: AZD2936

INTERVENTIONS:
Drug: AZD2936 — Anti-TIGIT/Anti-PD-1 Bispecific Antibody
  Other Names: Rilvegostomig

SUMMARY:
This is a Phase I/II study designed to evaluate if experimental anti-TIGIT/anti-PD-1 bispecific antibody rilvegostomig (AZD2936) is safe, tolerable and efficacious in participants with Advanced or Metastatic Non-small Cell Lung Cancer.

DETAILED DESCRIPTION:
This is a first-time-in-human (FTIH), open-label, multicenter, multi-part, dose-escalation and dose-expansion study to evaluate the safety, pharmacokinetics (PK), pharmacodynamics, and efficacy of rilvegostomig (AZD2936) in adult participants with stage III unresectable or stage IV NSCLC. The study includes 4 parts: Part A (dose escalation) and Parts B-E (dose expansion).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Aged 18 or above
* Part A and Part B: Unresectable stage III or stage IV squamous or non-squamous NSCLC not amenable to curative surgery or radiation. Part C and Part D: Stage IV squamous or non-squamous NSCLC not amenable to curative surgery or radiation. Part E: Stage IV squamous NSCLC not amenable to curative surgery or radiation.
* Documented PD-L1 expression by PD-L1 IHC per local report.
* Part A and Part B: Confirmed progression during treatment with a CPI-including regimen.
* Part C and Part D: No prior I/O treatment for metastatic NSCLC.
* Part E: No prior treatment for metastatic NSCLC.
* ECOG performance status of 0 or 1 at enrolment.
* Life expectancy of ≥ 12 weeks at enrolment.
* Have at least 1 measurable lesion per RECIST v1.1.
* Adequate bone marrow, liver and kidney function

Exclusion Criteria:

* Sensitizing epidermal growth factor receptor (EGFR) mutations or anaplastic lymphoma kinase (ALK) fusion
* Documented test result for any other known genomic alteration for which a targeted therapy is approved in first line per local standard of care (e.g. ROS1, NTRK fusions, BRAF, V600E mutation)
* Previous treatment with an anti-TIGIT therapy
* Any concurrent chemotherapy, radiotherapy, investigational, biologic, or hormonal therapy for cancer treatment.
* Part A and Part B: Primary or secondary resistance after treatment with 2 or more regiments including a CPI.
* Part C and Part D: Any prior systemic treatment with an immune oncology agent (prior administration of immune-oncology agent for curative intent to treat other invasive malignancy is permitted).

Treatment with one previous systemic chemotherapy will be allowed.

* Part E: Any prior systemic treatment for metastatic NSCLC, including but not limited to chemotherapy, anti-PD-1, anti-PD-L1, anti-CTLA-4.
* Symptomatic central nervous system (CNS) metastasis.
* Thromboembolic event within 3 months prior to enrolment.
* Other invasive malignancy within 2 years prior to screening.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2026-08-18 (Estimated); Study Completion 2028-03-16 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with adverse events (AEs) and immune mediated AEs (imAEs), serious AEs (SAEs), dose limiting toxicities (DLTs), vital signs, and abnormal laboratory parameters | Part A, B, C, D and E: From the time of informed consent until 90 days after the last dose of rilvegostomig
  A DLT is a toxicity defined by the study protocol that occurs from the first dose of study intervention up to the end of the DLT evaluation period that is assessed as clearly unrelated to the primary disease or intercurrent illness.
Rate of rilvegostomig discontinuation due to toxicity | Part A, B, C, D and E: From first dose to the last dose of rilvegostomig (an average of 6 months)
  Percentage of participants with AEs leading to discontinuation of rilvegostomig
Objective Response Rate (ORR) | Part B, C, D and E: From first dose of rilvegostomig to progressive disease (PD) or death in the absence of disease progression (approximately 2 years)
  Percentage of participants with a confirmed Complete Response (CR) or Partial Response (PR) according to RECIST v1.1

SECONDARY OUTCOMES:
ORR | Part A: From first dose of rilvegostomig to PD or death in the absence of disease progression (approximately 2 years).
  Percentage of participants with a confirmed CR or PR according to RECIST v1.1
Disease control rate (DCR) | Part A, B, C, E: From first dose of rilvegostomig to PD or death in the absence of disease progression (approximately 2 years). Part D: From randomization to PD or death in the absence of disease progression (approximately 2 years).
  Percentage of participants who have a best objective response of confirmed CR or PR or who have SD lasting for at least a certain time of period after start of treatment
Duration of response (DoR) | Part A, B, C, D and E: From first dose of rilvegostomig to PD or death in the absence of disease progression (approximately 2 years).
  The time from first response according to RECIST v1.1 until progression or death in the absence of disease progression
Durable response rate (DRR) | Part A, B, C, D and E: From first dose of rilvegostomig to PD or death in the absence of disease progression (approximately 2 years).
  The percentage of participants according to RECIST v1.1 with a confirmed CR or PR lasting 6 months or more
Progression-free survival (PFS) | Part B, C, E: From first dose of rilvegostomig to PD or death in the absence of disease progression (approximately 2 years). Part D: From randomization to PD or death in the absence of disease progression (approximately 2 years).
  The time from first dose of study intervention until the date of objective disease progression or death in the absence of disease progression
Measure the receptor occupancy (RO) of TIGIT and PD-1 on peripheral blood | Part A, B: From first dose of study intervention, at predefined intervals throughout the administration of rilvegostomig (approximately 2 years). The predefined intervals for Part A will be different from Part B.
  Evaluation of the target engagement of rilvegostomig in peripheral blood
PK of rilvegostomig: Maximum plasma concentration of the study drug (Cmax) | From first dose of study intervention, at predefined intervals throughout the administration of rilvegostomig (approximately 2 years). The predefined intervals for Part A will be different from Part B, C, D and E.
  Maximum observed plasma concentration of rilvegostomig
PK of rilvegostomig: Area under the concentration-time curve (AUC) | From first dose of study intervention, at predefined intervals throughout the administration of rilvegostomig (approximately 2 years). The predefined intervals for Part A will be different from Part B, C, D and E.
  Area under the plasma concentration-time curve
PK of rilvegostomig: Clearance | From first dose of study intervention, at predefined intervals throughout the administration of rilvegostomig (approximately 2 years). The predefined intervals for Part A will be different from Part B, C, D and E.
  A pharmacokinetic measurement of the volume of plasma from which the study intervention is completely removed per unit time.
PK of rilvegostomig: Terminal elimination half-life (t 1/2) | From first dose of study intervention, at predefined intervals throughout the administration of rilvegostomig (approximately 2 years). The predefined intervals for Part A will be different from Part B, C, D and E.
  Terminal elimination half life
Incidence of anti-drug antibodies (ADA) against rilvegostomig in serum | From first dose of study intervention, at predefined intervals throughout the administration of rilvegostomig (approximately 2 years). The predefined intervals for Part A will be different from Part B, C, D and E.
  Immunogenicity of rilvegostomig

CONTACTS AND LOCATIONS:
Locations (43):
- United States (6):
  - Research Site, Orange, California
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Rochester, Minnesota
  - Research Site, Houston, Texas
  - Research Site, Fairfax, Virginia
- Research Site, Melbourne, Australia
- Belgium (2):
  - Research Site, Anderlecht
  - Research Site, Leuven
- Brazil (5):
  - Research Site, Florianópolis
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- China (3):
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Wuhan
- Research Site, Copenhagen, Denmark
- France (2):
  - Research Site, Dijon
  - Research Site, Toulouse
- Research Site, Tbilisi, Georgia
- Japan (4):
  - Research Site, Kashiwa
  - Research Site, Niigata
  - Research Site, Sendai
  - Research Site, Tokyo
- Malaysia (2):
  - Research Site, Kuala Lumpur
  - Research Site, Kuching
- Research Site, Chisinau, Moldova
- Netherlands (3):
  - Research Site, Groningen
  - Research Site, Leiden
  - Research Site, Utrecht
- Research Site, Singapore, Singapore
- Research Site, Seoul, South Korea
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid
- Taiwan (3):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Chanthaburi
  - Research Site, Muang
- United Kingdom (2):
  - Research Site, Leicester
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level datain an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access.For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home